CLINICAL TRIAL: NCT00814931
Title: A Phase 1, Multiple Dose, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Examining the Effects of CXB722 in Mitigating Neuroendocrine Stress Response in Healthy Males
Brief Title: Examining the Effects of CXB722 in Neuroendocrine Stress Response in Healthy Males
Acronym: CXB722-100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CeNeRx BioPharma Inc. (Industry)
Responsible Party: Carlos Santana, MD, USF Physicians Group
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG0114
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Stress; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — pivagabine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment Group
  Interventions: Drug: CXB722
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CXB722 — 900 mg CXB722 oral liquid suspension twice a day for 8 days
  Other Names: Pivagabine
  Arms: 1
Drug: Placebo — matching oral liquid suspension placebo twice a day for 8 days
  Arms: 2

SUMMARY:
The purpose of this study is to assess the effects of CXB722 on neuroendocrine stress response and subjective reports related to mood and stress during and after experimentally induced stress among healthy young males.

DETAILED DESCRIPTION:
Acute stress produces a cascade of physiological and psychological effects, including increased cardiovascular function, increases in circulating levels of stress hormones and neurotransmitter levels, and changes in mood and subjective state. The Trier Social Stress Test (TSST) is a standardized, well-validated procedure that was developed in order to provide a controlled method for exposing subjects to a stressor. The TSST consists of a public speaking and a mental arithmetic test performed in the context of a mock job interview.

A drug that could safely block or mitigate the stress response would have multiple applications in medicine, beyond treating anxiety, because stress is associated with many disease states, including cardiovascular disease. The drug being studied, CXB722, is thought to show promise in diminishing the physiologic and psychological effects of stress.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18 to 34 years of age, inclusive, at screening
* Able to read, understand and converse in English
* Able to read, understand, and provide written, dated informed consent
* Willing to refrain from the use of any concomitant medications (including over-the counter (OTC)) and nutritional/herbal supplements and comply with all study requirements
* Willing to submit to daily breathalyzer testing each day study medication is administered over the course of the study
* In good general health as ascertained by medical history, physical examination (PE) including measurement of vital signs, clinical laboratory evaluations, and 12-lead electrocardiogram (ECG)

Exclusion Criteria:

* Evidence on physical examination or laboratory findings of chronic liver or renal disease or other chronic physical disorders
* Evidence of cardiovascular disease on 12 lead ECG, vital signs or laboratory findings
* Significant anxiety as indicated by a score of 47 or higher on the "Trait" score of Spielberger State-Trait Anxiety Scale
* Family history (first degree relative) of hypertension or cardiovascular disease prior to age 40
* Evidence on physical or laboratory examination of endocrinopathies or immunopathies, including HIV
* BMI of 30 or greater, evidence of significant recent weight change or history of obesity
* History of any psychiatric disorder, or evidence of such a disorder based on a psychiatric evaluation which includes the Structured Clinical Interview for DSM-IV-TR (SCID)
* History of any physical condition which, in the investigator's opinion, might put the participant at risk or interfere with the interpretation of study results
* Use of any prescription or over-the-counter (OTC) medications (including herbal remedies) within 14 days of study randomization
* Use of tobacco products or any nicotine-containing products (e.g., gum, patch) within the past 6 months (prior to screening)
* Positive screening urine test for nicotine or drugs of abuse: cannabinoids, cocaine, amphetamines, barbiturates, opiates, benzodiazepines, or alcohol in the blood
* Unwillingness to agree to avoid strenuous activity over the course of the study
* Poor likelihood, in the investigator's judgment, of full cooperation during the study and/or poor compliance is anticipated
* Previously screened for this trial
* Consumes more than four cups of coffee daily
* Deviates from normal nocturnal sleeping patterns

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Plasma cortisol and salivary cortisol levels | Screening and Study Day 8

SECONDARY OUTCOMES:
Plasma ACTH | Screening and Study Day 8
Plasma epinephrine and norepinephrine | Screening and Study Day 8
Profile of Mood States (POMS) Tension-Anxiety | Screening and Study Day 8
Fatigue-Inertia, and Vigor-Activity factor scores | Screening and Study Day 8
"State" score on the Spielberger State-Trait Anxiety Scale (SSTAS) | Screening and Study Day 8
Seven Visual Analog Scales (VAS) | Screening and Study Day 8
HR, and systolic and diastolic BP | Screening and Study Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Santana, MD, Principal Investigator — USF Physicians Group, Associate Professor, Director of Adult Outpatient Services, Department of Psychiatry and Behavioral Medicine
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Kirschbaum C, Strasburger CJ, Langkrar J. Attenuated cortisol response to psychological stress but not to CRH or ergometry in young habitual smokers. Pharmacol Biochem Behav. 1993 Mar;44(3):527-31. doi: 10.1016/0091-3057(93)90162-m. PMID 8451256